CLINICAL TRIAL: NCT05861102
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Jaktinib in Subjects With Active Ankylosing Spondylitis(AS)
Brief Title: Efficacy and Safety Study of Jaktinib in Subjects With Active Ankylosing Spondylitis(AS)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZGJAK029
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jaktinib 100mg BID (twice daily) (Experimental)
  Interventions: Drug: Jaktinib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jaktinib — Participants will receive 100 mg Jaktinib orally twice daily for 16 weeks
  Arms: Jaktinib 100mg BID (twice daily)
Drug: Placebo — Participants will receive matching placebo orally twice daily for 16 weeks
  Arms: Placebo

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, efficacy and safety study of Jaktinib in subjects with active Ankylosing Spondylitis(AS).

DETAILED DESCRIPTION:
Approximately 258 eligible subjects (129 per arm) will be randomized in a 1:1 ratio to Jaktinib 100mg BID (twice daily) or matching placebo BID for a total of 16 weeks of blinded treatment. During the 16-week treatment period subjects will visit the clinic every two weeks until the Week 4 visit and then every 4 weeks until the completion of Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to understand the study and signed the informed consent.
* 18-65 years, male or female.
* Participants with a clinical diagnosis of ankylosing spondylitis (AS), and radiologic evidence (x-ray) fulfilling the Modified New York criteria for AS(1984).
* Participants must have baseline disease activity as defined by having a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score ≥ 4 and a Patient's Assessment of Total Back Pain score ≥ 4 based on a 0 - 10 Numeric Rating Scale (NRS) at the Screening and Baseline Visits.
* Participants may be receiving the following Disease-Modifying Anti-Rheumatic Drugs(DMARDs) at the time of the screening visit. These medications should be continued throughout the entire study and doses should remain unchanged.
* Participants has had an inadequate response to at least two Nonsteroidal Anti-inflammatory Drugs (NSAIDs) over an at least 4-week period in total at maximum recommended or tolerated doses, or participant has an intolerance to or contraindication for NSAIDs.
* Participants who are regularly taking NSAIDs (including COX-1 or COX-2 inhibitors) as part of their AS therapy are required to be on a stable dose for at least 2 weeks before randomisation.
* Participants receiving non-prohibited concomitant medications for any reason must be willing to stay on a stable regimen as defined in the protocol.

Exclusion Criteria:

* History of known or suspected complete ankylosis of the spine.
* Any subject with condition affecting oral drug absorption.
* Participants taking high potency opioid analgesics (e.g. methadone, hydromorphone, morphine) within 4 weeks before randomization.
* Participants on any other DMARDs within 4 weeks or five half-lives (whichever is longer) of the drug prior to the Baseline visit.
* Participants has a history of inflammatory arthritis of different etiology other than axial SpA (including but not limited to rheumatoid arthritis, mixed connective tissue disease, systemic lupus erythematosus, reactive arthritis, scleroderma, polymyositis, dermatomyositis, fibromyalgia), or any arthritis with onset prior to 17 years of age.
* Significant trauma or surgery procedure within 8 weeks prior to randomization, or any planned elective surgery during the study period.
* Participants with a known immunodeficiency disorder or a first degree relative with a hereditary immunodeficiency.
* Participants with any condition possibly affecting oral drug absorption, eg, gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery.
* Use of any investigational drug and/or devices within 4 weeks of randomization or a period of 5 half-lives of the investigational drug, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Assessment in Ankylosing Spondylitis (ASAS) 40 response at Week 16 | Week 16
  ASAS40 is defined as a >= 40% improvement and an absolute improvement of ≥ 2 units (on a scale of 0 to 10) from Baseline in at least 3 of the 4 domains (patient's global assessment, back pain, function and inflammation) with no worsening at all in the remaining domain.

SECONDARY OUTCOMES:
Percentage of Participants with Assessment in Ankylosing Spondylitis (ASAS) 20 response at Week 16. | Week 16
  ASAS20 is defined as a >= 20% improvement and an absolute improvement of >= 1 units (on a scale of 0 to 10) from Baseline in at least 3 of the 4 domains (patient's global assessment, back pain, function and inflammation) with no deterioration in the remaining domain (where deterioration is defined as a worsening of >= 20% and a net worsening of >= 1 unit [on a scale of 0 to 10])
Percentage of Participants with Assessment in Ankylosing Spondylitis (ASAS) 40 response at Week 2、4、8 and 12. | Week 2、4、8 and 12
  ASAS40 is defined as a >= 40% improvement and an absolute improvement of ≥ 2 units (on a scale of 0 to 10) from Baseline in at least 3 of the 4 domains (patient's global assessment, back pain, function and inflammation) with no worsening at all in the remaining domain.
Percentage of Participants with Assessment in Ankylosing Spondylitis (ASAS) 20 response at Week 2、4、8 and 12. | Week 2、4、8 and 12
  ASAS20 is defined as a >= 20% improvement and an absolute improvement of >= 1 units (on a scale of 0 to 10) from Baseline in at least 3 of the 4 domains (patient's global assessment, back pain, function and inflammation) with no deterioration in the remaining domain (where deterioration is defined as a worsening of >= 20% and a net worsening of >= 1 unit [on a scale of 0 to 10])

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, Principal Investigator — RenJi Hospital
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China